CLINICAL TRIAL: NCT05429528
Title: Evaluating A Promising Food Policy Intervention Using NUSMart: A Sin-Tax Scheme
Brief Title: Understanding Food Choices in Saudi Arabia- Taxes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: World Bank (Other); Public Health Authority of Saudi Arabia (Unknown)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 7202186
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diet, Healthy
Keywords: Implicit/ Explicit Tax; Sugar-sweetened beverages tax; Diet quality; Online grocery shopping; Kingdom of Saudi Arabia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Arm 1) (No Intervention): Participants will experience a default version of NUSMart which replicates the traditional shopping experience of online grocery stores with no FOP labels.
- Implicit Tax Arm (Arm 2) (Experimental): Similar to Arm 1 except that an implicit tax is levied on qualifying beverages.
  Interventions: Behavioral: Implicit Tax
- Explicit Tiered Tax Arm (Arm 3) (Experimental): Similar to Arm 1 except that an explicit tiered tax is levied on qualifying food and beverage products.
  Interventions: Behavioral: Explicit Tiered Tax

INTERVENTIONS:
Behavioral: Implicit Tax — This will be levied only on certain beverage categories: a 50% tax on the sales prices of carbonated drinks and sugar-sweetened beverages (SSBs) and 100% tax on the sales prices of energy drinks (milk, milk-based products, and natural fruit juice are excluded).
  Arms: Implicit Tax Arm (Arm 2)
Behavioral: Explicit Tiered Tax — This is an explicit tiered tax based on (underlying) Nutri-Score (NS) grades which will be levied on all food and beverages. In this arm, the investigators implement a 20% sales tax on the retail price for NS D beverages and 10% for NS D foods along with a 50% sales tax on NS E beverages and 20% on NS E foods. The NS labels will not be displayed.
  Arms: Explicit Tiered Tax Arm (Arm 3)

SUMMARY:
Using a 3-arm randomized controlled trial, the investigators aim to rigorously evaluate the effects of two different taxation policies on diet quality. The first is an implicit sales tax that will be levied only on beverages in a manner that mirrors the current Kingdom of Saudi Arabia (KSA) beverage taxes and the second is an explicit Nutri-Score (NS) based tiered tax that is levied on all food and beverage products. The investigators will use an experimental online grocery store, called NUSMart, which is similar in design to commercial web-based grocery stores to test these two taxation policies. Participants will be randomly assigned to one of the following arms and asked to complete a one-time hypothetical shop.

Arm 1 (Control): Participants will experience a default version of NUSMart which replicates the traditional shopping experience of online grocery stores with no FOP labels.

Arm 2 (Implicit Tax): Same as Arm 1 NUSMart except that an implicit tax will be levied only on beverages: a 50% sales tax on carbonated drinks and sugar-sweetened beverages (SSBs) and 100% tax on energy drinks (milk, milk-based products, and natural fruit juice are excluded).

Arm 3 (Explicit Tiered Tax): Same as Arm 1 NUSMart except that an explicit tiered tax based on (underlying) NS is levied on (sale price of) all food and beverages. NS assesses overall nutritional quality of products on the basis of 7 nutrients (calories, saturated fats, sugar, salt, fiber, protein and percentage of fruits, vegetables and nuts) from A to E (best to worst). In this arm, the investigators implement a 20% sales tax on the retail price for NS D beverages and 10% for NS D foods along with a 50% sales tax on NS E beverages and 20% on NS E foods.

The investigators hypothesize the following:

Hypothesis 1: Diet quality of food purchases, measured by the weighted average Nutri-Score point, will be highest in the explicit tiered tax arm, followed by the implicit tax arm, followed by the control.

Hypothesis 2: Average calories, sugar, sodium, and saturated fat per serving will be lowest in the explicit tiered tax arm, followed by the implicit tax arm, followed by the control.

DETAILED DESCRIPTION:
Experimental design & procedures

The aim of this study is to use a 3-arm randomized controlled trial with an online grocery store known as NUSMart, to rigorously evaluate the effect of two different taxation policies i.e., implicit tax on select beverages and an explicit tiered tax on all products, on diet quality.

1. Tax Strategies

   The investigators tested 2 different types of taxation strategies in this study. They are as follows:
   1. Implicit Tax: This will be levied only on certain beverage categories: a 50% sales tax on carbonated drinks and sugar-sweetened beverages (SSBs) and 100% tax on energy drinks (milk, milk-based products, and natural fruit juice are excluded).
   2. Explicit Tiered Tax: This is an explicit tiered tax based on (underlying) Nutri-Score (NS) grades which will be levied on all food and beverages. In this arm, the investigators implement a 20% sales tax on the retail price for NS D beverages and 10% for NS D foods along with a 50% sales tax on NS E beverages and 20% on NS E foods. The NS labels will not be displayed.
2. Overview of RCT Design

   To test these labels, the investigators used three different versions of NUSMart. Each participant was randomly assigned to one of the following arms and asked to complete a one-time hypothetical shop.

   Arm 1: Control arm. Participants experience an unmodified version of NUSMart, which replicates the traditional shopping experience of online grocery stores.

   Arm 2: Similar to Arm 1 except that an implicit tax is levied on qualifying beverages.

   Arm 3: Similar to Arm 1 except that an explicit tiered tax is levied on qualifying food and beverage products.

   To minimize hypothetical shopping biases, the investigators set a minimum spending value per person per week and adjusted the total minimum spending value depending on household size. Additionally, participants will have to shop from 4 different NUSMart categories and purchase at least one beverage product to be able to successfully checkout their cart. Finally, participants will be told that there is up to a 50% probability that they will be asked to actually purchase the items in their final checked-out cart when in reality they will never be asked to make any purchase.
3. Subject related procedures

As the investigators have done in prior studies, participants will be recruited if they are KSA residents aged 18 years or older, can speak Arabic and are primary weekly shoppers for their households. Recruitment will be done through Facebook advertisements boosted using an automation tool called Revealbot to help optimise workflow.

On recruitment, they will be asked to fill in a baseline questionnaire to collect demographic and health characteristics, which should take approximately 10-15 minutes to complete. The baseline questionnaire includes a question as to whether any household members have a medical condition, such as diabetes or hypertension, which requires limiting the types of foods they eat. Investigators ask this question to allow for testing whether the interventions differentially influence these households, with the expectation that households with less healthy patients may obtain greater benefits from purchasing baskets with higher mean Nutri-Scores. Since the objective of this randomized control trail (RCT) is to quantify the effectiveness of the interventions on diet quality, a precursor to NCDs, the collection of household health indicators is reasonable.

Upon completion of the baseline survey, participants will be randomly assigned to one of the 3 shopping conditions (Arm 1 [Control], Arm 2, or Arm 3) and redirected to NUSMart to log in and begin shopping immediately.

On NUSMart, they will be asked to purchase their weekly groceries with a minimum spend of SAR 75 (equivalent to 20 USD) per person per week (the total minimum spending value will depend on the household size). Each participant will therefore shop only once during the study in one of the arms (1, 2 or 3) which will be randomly assigned to them.

Participants will be given explicit instructions to purchase groceries for the purposes of breakfast, lunch, dinner, snacks, and beverage consumption for one week keeping in mind that they will not be consuming any meals outside. The stores will be set up such that participants will not be allowed to check out with their cart unless they have selected items from 4 different NUSMart categories and purchase at least one beverage. This is to ensure that participants shop as though they are shopping for their own consumption i.e., to minimize hypothetical biases. As mentioned earlier, participants will be reminded that there is up to a 50% probability that they will be asked to actually purchase the products in the final cart they check out from the store.

A post-study survey will be conducted after the shop to collect participant opinions on the labels and understand their impact better.

ELIGIBILITY:
Inclusion Criteria:

* People who are KSA (Kingdom of Saudi Arabia) citizens
* Age of 18 and above,
* Arabic speakers, and
* A weekly primary grocery shopper for their households can participate in this study.

Exclusion Criteria:

* People who are not KSA citizens,
* Under 18 years of age,
* Cannot speak Arabic, or
* Are not weekly primary grocery shoppers for their households cannot participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2490 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Value of Nutri-Score | After completion of data collection, an average of about 5 months
  Diet quality measured by the weighted (by the number of servings) average of all purchased products' Nutri-Score for the shopping trip. Nutri-Score is a holistic dietary index based on the British Food Standard Agency Nutrient Profiling System that grades food and beverage products from A to E where A indicates the highest nutritional quality and E indicates the lowest nutritional quality.

SECONDARY OUTCOMES:
Quantity of other Nutrients | After completion of data collection, an average of about 5 months
  calories per serving, grams of sugars per serving, milligrams of sodium per serving, grams of saturated fat per serving.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No